CLINICAL TRIAL: NCT05230862
Title: Does a Multi-ingredient Pre-workout Supplement Enhance Cycling Time Trial
Brief Title: Does a Multi-ingredient Pre-workout Supplement Enhance Cycling Time Trial Performance?
Acronym: MIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: OpenFit LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-M-38
Record Dates: First submitted 2022-01-10; First posted 2022-02-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ladder Supplement (Experimental): Ladder Supplement
  Interventions: Dietary Supplement: Ladder Supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ladder Supplement — Caffeine 200mg L-Theanine 200mg L-Citrulline 6g Creatine 5g Beta-Alanine 1.6g Phosphatidylserine 100mg
  Arms: Ladder Supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the present study is to test the effect of ingesting a multi-ingredient pre- exercise supplement containing caffeine, creatine, beta-alanine and L-Citrulline compared to a placebo, on endurance exercise performance.

ELIGIBILITY:
Exclusion criteria:

* Any diagnosed metabolic health condition
* Pregnant
* Non-habitual caffeine intake
* Smoker
* No endurance training
* Diagnosed Cardiovascular disease
* Recent history of musculoskeletal injury
* Anti-depressant and anti-anxiety medication

Inclusion criteria

* Age 18-40
* Healthy
* Highly trained endurance athletes (V̇O2max: males >55 and females >50 mL⋅kg bm-1⋅min-1)
* Both males and females are allowed to participate. If females are on the oral contraceptive pill they are to be tested on consecutive weeks. If they are not on the oral contraceptive pill, then female subjects are to be tested every 4 weeks, at the same point of their menstrual cycle.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise Performance | 15 Minitues
  Work done during 15 min time trial (TT)

SECONDARY OUTCOMES:
Alertness | 1 Hour
  Visual analog scale
Motivation | 1 Hour
  Visual analog scale
Rate of perceived exertion | 1 Hour
  Visual analog scale
Gas analysis | 1 Hour
  Analysis of expired gas

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport and Health Sciences, Exeter, United Kingdom